CLINICAL TRIAL: NCT02828930
Title: A Single-Center, Open-Label Study Investigating the Excretion Balance, Pharmacokinetics, Metabolism, and Absolute Oral Bioavailability of a Single Oral Dose of [14C]-Labeled Idasanutlin and an Intravenous Tracer Dose of [13C]-Labeled Idasanutlin in a Single Cohort of Patients With Solid Tumors
Brief Title: A Study to Determine the Excretion Balance, Pharmacokinetics, Metabolism and Absolute Oral Bioavailability of a Single Oral Dose of [14C]-Labeled Idasanutlin and an Intravenous Tracer Dose of [13C]-Labeled Idasanutlin in a Single Cohort of Participants With Solid Tumors (Malignancies)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NP29910; RG7388 (Other: Roche); 2015-002532-40 (EudraCT Number)
Record Dates: First submitted 2016-07-07; First posted 2016-07-12 (Estimated); Last update posted 2017-12-18 (Actual); Status verified 2017-12

CONDITIONS: Solid Tumors
MeSH Terms: interventions — RG7388

ARMS (1):
- Idasanutlin (Experimental): On Day 1, 300 milligram (mg) idasanutlin tablet orally and 100 mg [14C]-radiolabeled idasanutlin capsule orally (2, 50 mg capsules containing approximately 100 microcurie of radioactivity). After 5 hours and 45 minutes of the oral dose, 100 microgram (mcg) of [13C]-radiolabeled idasanutlin will be administered over a 15-minute intravenous (IV) infusion. On Day 11, idasanutlin matching placebo aqueous dispersion orally and approximately after 1 hour, 400 mg idasanutlin tablet will be administered orally in the form of an aqueous dispersion. On Day 19, 400 mg idasanutlin tablet will be administered orally in the form of an aqueous dispersion. Participants, who are eligible to enter in optional treatment extension phase, will continue treatment with idasanutlin 200 mg tablet orally once daily for 5 days, and no treatment during 23 days of 28-day cycle, until the development of progressive disease, unacceptable toxicity, consent withdrawal or any other criteria for removal.
  Interventions: Drug: Idasanutlin; Drug: Placebo; Drug: [13C]-radiolabeled Idasanutlin; Drug: [14C]-radiolabeled Idasanutlin

INTERVENTIONS:
Drug: Idasanutlin — Idasanutlin 300 mg tablet orally on Day 1; 400 mg tablet orally on Day 11 and Day 19. Participants, who are eligible to enter in optional treatment extension phase, will continue treatment with idasanutlin 200 mg tablet orally once daily for 5 days of 28-day cycle.
  Other Names: RO5503781
Drug: Placebo — Placebo matching to idasanutlin aqueous dispersion will be administered orally on Day 11.
Drug: [13C]-radiolabeled Idasanutlin — [13C]-radiolabeled idasanutlin 100 mcg will be administered as IV infusion over 15-minute on Day 1.
Drug: [14C]-radiolabeled Idasanutlin — [14C]-radiolabeled idasanutlin 100 mg capsule (2, 50 mg capsules containing approximately 100 microcurie of radioactivity) will be administered orally on Day 1.

SUMMARY:
The purpose of this single-center, open-label, non-randomized study is to assess the excretion balance, pharmacokinetics, metabolism and absolute oral bioavailability of [14C]-labeled idasanutlin administered orally and [13C]-labeled idasanutlin administered intravenously in a single cohort of eligible participants. Participants will be screened for participation in this study within 21 days of receiving the first dose of study drug on Day 1. Treatment period will continue up to Day 28 after which participants will enter 28 day follow-up or the optional treatment extension of idasanutlin, depending on safety parameters and as per opinion of the Investigator.

ELIGIBILITY:
Inclusion Criteria:

* Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 2, at the discretion of the Investigator
* Histologically or cytologically confirmed advanced malignancy, except leukemia and lymphoma
* Measureable or evaluable disease by Response evaluation criteria in solid tumors (RECIST) version 1.1, with no more than a single active malignancy in the previous 3 to 5 years prior to the administration of study drug
* Life expectancy of at least 12 weeks
* Participants taking opioid analgesics for pain should be on a stable pain and palliative care bowel regimen for one month prior to the first dose of study medication
* Adequate bone marrow, hepatic, and renal function
* Agreement to remain abstinent or use contraceptive methods specified in the study

Exclusion Criteria:

* History of any form of leukemia, except for Stage 0 - 1 chronic lymphocytic leukemia, not requiring treatment in addition to their underlying malignancy
* Have received hormonal therapy within the two weeks prior to the first dose of study drug
* Have pre-existing gastrointestinal disorders that may interfere with proper absorption of the drug
* History of seizure disorders or unstable Central Nervous System metastases (participants with stable CNS metastases allowed)
* Have any severe and/or uncontrolled medical conditions or other conditions that could affect their participation in the study
* Receive certain per protocol prohibited medications while on study. These medications must be discontinued 7 days prior to start of study drug
* Have bone marrow disorders, electrolyte imbalance, infrequent bowel movements (less than once per 48 hours), coagulopathy, platelet disorder or history of non-drug induced thrombocytopenia
* Positive for human immunodeficiency virus currently receiving combination anti-retroviral therapy
* Regular work with ionizing radiation or radioactive material or treated with radiotherapy within 3 weeks prior to the first dose of study drug
* Refuse to potentially receive blood products and/or have a hypersensitivity to blood products

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2016-09-08 (Actual); Primary Completion 2017-06-19 (Actual); Study Completion 2017-06-19 (Actual)

PRIMARY OUTCOMES:
Time to Reach Maximum Observed Plasma Concentration (Tmax) of Unlabeled Idasanutlin | 0 Hour (hr) predose, 1, 3, 6, 7, 24, 48, 96, 120, 144, 240 hrs postdose
Maximum Observed Plasma Concentration (Cmax) of Unlabeled Idasanutlin | 0 hr predose, 1, 3, 6, 7, 24, 48, 96, 120, 144, 240 hrs postdose
Area Under the Plasma Concentration Time-Curve From Time Zero to Extrapolated Infinite Time (AUC [0-inf]) of Unlabeled Idasanutlin | 0 hr predose, 1, 3, 6, 7, 24, 48, 96, 120, 144, 240 hrs postdose
Area Under the Plasma Concentration Time-Curve From Zero to the Last Measured Concentration (AUC[0-last]) of Unlabeled Idasanutlin | 0 hr predose, 1, 3, 6, 7, 24, 48, 96, 120, 144, 240 hrs postdose
Plasma Elimination Half-Life (t1/2) of Unlabeled Idasanutlin | 0 hr predose, 1, 3, 6, 7, 24, 48, 96, 120, 144, 240 hrs postdose
Plasma Apparent Elimination Rate Constant of Unlabeled Idasanutlin | 0 hr predose, 1, 3, 6, 7, 24, 48, 96, 120, 144, 240 hrs postdose
Apparent Oral Clearance (CL/F) of Unlabeled Idasanutlin | 0 hr predose, 1, 3, 6, 7, 24, 48, 96, 120, 144, 240 hrs postdose
Renal Clearance (CLr) of Unlabeled Idasanutlin | 0 hr predose, 1, 3, 6, 7, 24, 48, 96, 120, 144, 240 hrs postdose
Apparent Volume of Distribution (Vz/F) of Unlabeled Idasanutlin | 0 hr predose, 1, 3, 6, 7, 24, 48, 96, 120, 144, 240 hrs postdose
Cumulative Amount Excreted in Urine of Unlabeled Idasanutlin | 0 hr (within 24 hrs of dosing), pooled sample collected over time interval: 0-6, 6-12, 12-24, 24-48, 48-72, 72-96, 96-120, 120-144, 144-168, 168-192, 192-216, 216-240, 240-264 hrs postdose
Cumulative Amount Excreted in Feces of Unlabeled Idasanutlin | 0 hr (within 24 hrs of dosing), pooled sample collected over time interval: 0-6, 6-12, 12-24, 24-48, 48-72, 72-96, 96-120, 120-144, 144-168, 168-192, 192-216, 216-240, 240-264 hrs postdose
Tmax of Idasanutlin Metabolite | 0 hr predose, 1, 3, 6, 7, 24, 48, 96, 120, 144, 240 hrs postdose
Cmax of Idasanutlin Metabolite | 0 hr predose, 1, 3, 6, 7, 24, 48, 96, 120, 144, 240 hrs postdose
AUC (0-inf) of Idasanutlin Metabolite | 0 hr predose, 1, 3, 6, 7, 24, 48, 96, 120, 144, 240 hrs postdose
AUC(0-last) of Idasanutlin Metabolite | 0 hr predose, 1, 3, 6, 7, 24, 48, 96, 120, 144, 240 hrs postdose
Plasma t1/2 of Idasanutlin Metabolite | 0 hr predose, 1, 3, 6, 7, 24, 48, 96, 120, 144, 240 hrs postdose
Plasma Apparent Elimination Rate Constant of Idasanutlin Metabolite | 0 hr predose, 1, 3, 6, 7, 24, 48, 96, 120, 144, 240 hrs postdose
CL/F of Idasanutlin Metabolite | 0 hr predose, 1, 3, 6, 7, 24, 48, 96, 120, 144, 240 hrs postdose
CLr of Idasanutlin Metabolite | 0 hr predose, 1, 3, 6, 7, 24, 48, 96, 120, 144, 240 hrs postdose
Vz/F of Idasanutlin Metabolite | 0 hr predose, 1, 3, 6, 7, 24, 48, 96, 120, 144, 240 hrs postdose
Cumulative Amount Excreted in Urine of Idasanutlin Metabolite | 0 hr (within 24 hrs of dosing), pooled sample collected over time interval: 0-6, 6-12, 12-24, 24-48, 48-72, 72-96, 96-120, 120-144, 144-168, 168-192, 192-216, 216-240, 240-264 hrs postdose
Cumulative Amount Excreted in Feces of Idasanutlin Metabolite | 0 hr (within 24 hrs of dosing), pooled sample collected over time interval: 0-6, 6-12, 12-24, 24-48, 48-72, 72-96, 96-120, 120-144, 144-168, 168-192, 192-216, 216-240, 240-264 hrs postdose
Tmax of [13C]-Labeled Idasanutlin | 0 hr predose, 5hr 55 minutes (min), 6hr, 6hr 5min, 6hr 10min, 6hr 15min, 6hr 30min, 7, 10, 24, 48, 96, 120, 144, 240 hrs postdose
Cmax of [13C]-Labeled Idasanutlin | 0 hr predose, 5hr 55 min, 6hr, 6hr 5min, 6hr 10min, 6hr 15min, 6hr 30min, 7, 10, 24, 48, 96, 120, 144, 240 hrs postdose
AUC(0-inf) of [13C]-Labeled Idasanutlin | 0 hr predose, 5hr 55 min, 6hr, 6hr 5min, 6hr 10min, 6hr 15min, 6hr 30min, 7, 10, 24, 48, 96, 120, 144, 240 hrs postdose
AUC(0-last) of [13C]-Labeled Idasanutlin | 0 hr predose, 5hr 55min, 6hr, 6hr 5min, 6hr 10min, 6hr 15min, 6hr 30min, 7, 10, 24, 48, 96, 120, 144, 240 hrs postdose
Plasma t1/2 of [13C]-Labeled Idasanutlin | 0 hr predose, 5hr 55min, 6hr, 6hr 5min, 6hr 10min, 6hr 15min, 6hr 30min, 7, 10, 24, 48, 96, 120, 144, 240 hrs postdose
Absolute Oral Bioavailability of [13C]-Labeled Idasanutlin | Oral administration: 0 hr predose, 1, 3, 6, 7, 24, 48, 96, 120, 144, 240 hrs postdose; IV administration: 0 hr predose, 5hr 55min, 6hr, 6hr 5min, 6hr 10min, 6hr 15min, 6hr 30min, 7, 10, 24, 48, 96, 120, 144, 240 hrs postdose
Whole Blood and Plasma Cmax of [14C]-Labeled Idasanutlin | 0 hr predose, 1, 3, 6, 7, 24, 48, 96, 120, 144, 240 hrs postdose
Whole Blood and Plasma AUC(0-inf) of [14C]-Labeled Idasanutlin | 0 hr predose, 1, 3, 6, 7, 24, 48, 96, 120, 144, 240 hrs postdose0 hr predose, 1, 3, 6, 7, 24, 48, 96, 120, 144, 240 hrs postdose
Whole Blood and Plasma AUC(0-last) of [14C]-Labeled Idasanutlin | 0 hr predose, 1, 3, 6, 7, 24, 48, 96, 120, 144, 240 hrs postdose
Whole Blood and Plasma Apparent Elimination Rate Constant of [14C]-Labeled Idasanutlin | 0 hr predose, 1, 3, 6, 7, 24, 48, 96, 120, 144, 240 hrs postdose
Cumulative Amount of Radioactivity Excreted in Urine as Percentage of Dosed Radioactivity of [14C]-Labeled Idasanutlin | 0 hr (within 24 hrs of dosing), pooled sample collected over time interval: 0-6, 6-12, 12-24, 24-48, 48-72, 72-96, 96-120, 120-144, 144-168, 168-192, 192-216, 216-240, 240-264 hrs postdose
Cumulative Amount of Radioactivity Excreted in Feces as Percentage of Dosed Radioactivity of [14C]-Labeled Idasanutlin | 0 hr (within 24 hrs of dosing), pooled sample collected over time interval: 0-6, 6-12, 12-24, 24-48, 48-72, 72-96, 96-120, 120-144, 144-168, 168-192, 192-216, 216-240, 240-264 hrs postdose
CL/F of [13C]-Labeled Idasanutlin | 0 hr predose, 5hr 55min, 6hr, 6hr 5min, 6hr 10min, 6hr 15min, 6hr 30min, 7, 10, 24, 48, 96, 120, 144, 240 hrs postdose
Vz/F of [13C]-Labeled Idasanutlin | 0 hr predose, 5hr 55min, 6hr, 6hr 5min, 6hr 10min, 6hr 15min, 6hr 30min, 7, 10, 24, 48, 96, 120, 144, 240 hrs postdose
Whole Blood and Plasma Tmax of [14C]-Labeled Idasanutlin | 0 hr predose, 1, 3, 6, 7, 24, 48, 96, 120, 144, 240 hrs postdose
Cumulative Amount of Radioactivity Excreted in Feces on Toilet Tissue as Percentage of Dosed Radioactivity of [14C]-Labeled Idasanutlin | 0 hr (within 24 hrs of dosing), pooled sample collected over time interval: 0-6, 6-12, 12-24, 24-48, 48-72, 72-96, 96-120, 120-144, 144-168, 168-192, 192-216, 216-240, 240-264 hrs postdose

SECONDARY OUTCOMES:
Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs) | Baseline through 28 days after the last dose of study drug (maximum up to approximately 76 days)
Palatability Assessment Questionnaire Score for Aqueous Dispersion of Idasanutlin | 0 hr (pre-Day 11-dose), 0.5 hr, 1 hr, 1.5 hr, 2 hr, and 3 hr post-Day 11-dose
Aftertaste Survey Questionnaire Score for Aqueous Dispersion of Idasanutlin | 0 hr (pre-Day 11-dose), 0.5 hr, 1 hr, 1.5 hr, 2 hr, and 3 hr post-Day 11-dose

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (1):
- Magyar Honvedseg Egeszsegugyi Kozpont, Budapest, Hungary